CLINICAL TRIAL: NCT03206281
Title: Tall Stature Women Fetal Weight Estimation,Clinical Versus Sonographic Estimation
Brief Title: Tall Stature Women Fetal Weight Estimation
Acronym: TSFW
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Yair Daykan, Principal Investigator, M.D, Meir Medical Center
Other Study IDs: MMC-0016-17
Record Dates: First submitted 2017-06-20; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Ultrasonography, Prenatal
Keywords: clinical weight estimation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical fetal weight estimation: The fetal weight estimation will be taken by professional obstetrician durin her 39 week
  Interventions: Diagnostic Test: Fetal wight estimation
- Sonographic fetal weight estimation: The fetal weight estimation will be taken by professional Sonographic obstetrician durin her 39 week
  Interventions: Diagnostic Test: Fetal wight estimation

INTERVENTIONS:
Diagnostic Test: Fetal wight estimation — We will estimate the fetal weight by sonographic and clinical estimation

SUMMARY:
To investigate the difference of clinical VS sonographic fetal weight estimation of tall women stature (above 10t percentile)

DETAILED DESCRIPTION:
Women undergoing delivery after week 39 will be estimated of their fetal wight with clinical estimation and then sonographic estimation.

each women will be case control 1:1 for the actual fetal weight of the delivery.

the fetal weight will be blinded for each estimation.

Primary outcome is the actual fetal weight Secondary outcomes will be mode of delivery, fetal complication as APGAR score and fetal hypoxia and maternal complication as perineal laceration

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women above 172 cm height
* above 39 weeks of gestation

Exclusion Criteria:

* contraindication for vaginal delivery
* Intrauterus growth restriction

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women obove 172 cm hight
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-05 (Estimated); Primary Completion 2018-08-29 (Estimated); Study Completion 2018-09-29 (Estimated)

PRIMARY OUTCOMES:
The accuracy of fetal weight estimation | 2 weeks
  Comparing the sonographic and clinical fetal weight estimation to the actual fetal weight

SECONDARY OUTCOMES:
Mode of delivery and fetal complication | 2 weeks
  Vaginal Versus cesarian section delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Yes
within 6m of finishing the study

REFERENCES:
- [Derived] Daykan Y, Shavit M, Yagur Y, Schreiber H, Weitzner O, Schonman R, Biron-Shental T, Markovitch O. Fetal weight estimation in tall women: is ultrasound more accurate than clinical assessment? A prospective trial. Arch Gynecol Obstet. 2022 Mar;305(3):567-572. doi: 10.1007/s00404-021-06177-6. Epub 2021 Aug 11. PMID 34382135